CLINICAL TRIAL: NCT00855504
Title: Role of Cytokines in Association Between Periodontitis and Preeclampsia During Pregnancy
Brief Title: Association of Periodontitis and Preeclampsia During Pregnancy
Status: Completed | Type: Observational
Sponsor: Maulana Azad Medical College (Other)
Collaborators: University Grants Commission, New Delhi (Unknown)
Responsible Party: Principal Investigator, Ashok Kumar, Director Professor, Maulana Azad Medical College
Other Study IDs: 34-499/2008(SR)
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Preeclampsia; Periodontal Disease
Keywords: preeclampsia; periodontitis; cytokines
MeSH Terms: conditions — Pre-Eclampsia; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects: All the consecutive primigravidae who register in the antenatal clinic before 20 weeks of gestation

SUMMARY:
Infections affecting the mother during pregnancy may produce alterations in the normal cytokine and hormone-regulated gestation, which could result in preeclampsia, preterm labor, premature rupture of membranes, and preterm birth. Therefore, pregnant women with periodontal disease may show an alteration in the cytokine levels which may cause preeclampsia in them.

DETAILED DESCRIPTION:
The enrolled subjects will be evaluated on the basis of a pre-designed and pre-tested proforma with respect to history and clinical examination, obstetrics examination and ultrasonography. The periodontal examination consists of assessments at vestibular, lingual, mesial and distal sites of all present teeth.Five ml venous blood sample will be drawn from the patient at the time of enrollment before 20 weeks of gestation for the levels of cytokines (IL-4, IL-10, IFN-g and TNF-α. All the subjects will be followed- up till delivery. At the time of delivery, the details of pregnancy outcome (maternal and fetal) along with the measurement of the blood pressure will be recorded. A repeat of oral health evaluation will be done within 48 hours of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Singleton live pregnancy.
* Sure of her dates. (known dates of the last menstrual period)
* Age group 18-35 years.

Exclusion Criteria:

* Chronic hypertension
* Polyhydramnios
* Congenital malformation in fetus
* Diabetes
* Renal disease
* Cardiovascular disease
* Urolithiasis
* Parathyroid disease
* Systolic blood pressure measurement of more than 140mm Hg and diastolic blood pressure more than 90 mm Hg at first visit.
* Infections (bacterial vaginosis and chorioamnionitis)
* Antibiotic use during pregnancy
* Excessive body mass index
* Less than 20 natural teeth

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: primigravidae women with 14-20 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Association between preeclampsia and periodontal disease and its correlation with the variation in cytokine levels. | 3 years

SECONDARY OUTCOMES:
Correlation of relationship of periodontal disease with preeclampsia and pregnancy outcome. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Kumar, MD, Principal Investigator — Department of Obstetrics and Gynecology, Maulana Azad Medical College, New Delhi, India
Locations (1):
- Maulana Azad Medical College and Lok Nayak Hospital and Maulana Azad Institute of Dental Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Cota LO, Guimaraes AN, Costa JE, Lorentz TC, Costa FO. Association between maternal periodontitis and an increased risk of preeclampsia. J Periodontol. 2006 Dec;77(12):2063-9. doi: 10.1902/jop.2006.060061. PMID 17209792
- [Background] Contreras A, Herrera JA, Soto JE, Arce RM, Jaramillo A, Botero JE. Periodontitis is associated with preeclampsia in pregnant women. J Periodontol. 2006 Feb;77(2):182-8. doi: 10.1902/jop.2006.050020. PMID 16460242
- [Background] Canakci V, Canakci CF, Canakci H, Canakci E, Cicek Y, Ingec M, Ozgoz M, Demir T, Dilsiz A, Yagiz H. Periodontal disease as a risk factor for pre-eclampsia: a case control study. Aust N Z J Obstet Gynaecol. 2004 Dec;44(6):568-73. doi: 10.1111/j.1479-828X.2004.00323.x. PMID 15598299